CLINICAL TRIAL: NCT00461344
Title: A Multicenter, Open Label, Phase II Trial Evaluating Docetaxel + Anthracycline x 4 Cycles Followed by Docetaxel Single Agent x 4 Cycles as First-Line Therapy in Patients With Her2 Negative Locally Advanced or Metastatic Breast Cancer Who Have Relapsed ≥ 12 Months From Completion of Neoadjuvant/Adjuvant Taxotere®- Based Chemotherapy
Brief Title: Docetaxel + Doxorubicin as Neoadjuvant Chemotherapy in Patients With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to slow recruitment of patients
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976D_2504
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Ductal Carcinoma
Keywords: Breast
MeSH Terms: conditions — Carcinoma, Ductal | interventions — Docetaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Docetaxel
Drug: Doxorubicin

SUMMARY:
Primary: To determine the pathological remission following the chemotherapy combination docetaxel and doxorubicin in large breast cancer

Secondary:

* Clinical response rate
* To investigate the safety of docetaxel doxorubicin combination in the treatment for neoadjuvant chemotherapy of breast cancer
* Type of surgery (radical/conservative)

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified breast cancer
* Large (≥ 3 cm) breast cancer
* IIb-IIIa stage
* ECOG (Eastern Cooperative Oncology Group) status: 0-1-2
* Adequate bone marrow reserve: (Haemoglobin ≥ 12g/l, Absolute Neutrophil Count (ANC) ≥ 2.0x 10^9, Platelets ≥100 000)
* Laboratory results:
* Bilirubin ≤ Upper Limit Normal (ULN)
* Serum Glutamate Pyruvate Transaminase (SGPT) ≤ 2.5 ULN, Serum Glutamate Oxaloacetate Transaminase (SGOT) ≤ 2.5 ULN,
* Alk.phosph. ≤ 5.0 ULN,
* Creatinin ≤ ULN, if borderline calculated at ≤ 60ml/min
* Normal cardiac function (the result of Left Ventricular Ejection Function (LVEF) must be above the lower limit of normal for the institution)
* Negative pregnancy test
* Hormonal receptor status assessed

Exclusion Criteria:

* Pregnancy or lactation
* SGOT and/or SGPT > 1.5 upper limit normal, associated with Alk.phosph > 2.5 ULN
* Serious medical condition including but not limited to:
* Uncontrolled hypertension
* Active ulcus pepticum
* Non-stable diabetes mellitus
* Other contraindication of steroid treatment
* Myocardial infarction within the last 6 months prior study entry
* Significant neurologic/psychiatric disorders
* Active infection
* Peripheral neuropathy grade ≥ 2
* Unstable angina
* Severe arrhythmia
* Participation in other clinical trial
* Prior surgery, chemotherapy, hormonotherapy for breast cancer
* Past or current history of neoplasm other than breast cancer, except for: curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix, other cancer curatively treated and with no evidence of disease for at least 7 years
* History of hypersensitivity to the investigational products or to drugs with similar chemical structures
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol
* Treatment with any investigational product in the last 1 month before study entry.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-07; Primary Completion 2005-06 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Primary 1. to determine the pathological remission following the chemotherapy combination docetaxel and doxorubicin in large breast cancer

SECONDARY OUTCOMES:
Secondary: 1. Clinical response rate 2. to investigate the safety of docetaxel doxorubicin combination in the treatment for neoadjuvant chemotherapy of breast cancer 3. Type of surgery (radical/conservative)

CONTACTS AND LOCATIONS:
Overall Officials: László Erős, Study Director — sanofi-aventis Hungary